CLINICAL TRIAL: NCT05675683
Title: Real-World Assessment of Clinical Outcomes in Metastatic NSCLC Patients With MET Exon 14 Skipping Mutation and Brain Metastases Treated With Capmatinib
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC280AUS13
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Asymptomatic Brain Metastases: Patients with Asymptomatic Brain Metastases
  Interventions: Drug: Capmatinib
- Symptomatic Brain Metastases: Patient with Symptomatic Brain Metastases
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Capmatinib — Patients receiving Capmatinib

SUMMARY:
This was a retrospective, noninterventional cohort study of patients with a confirmed diagnosis of metastatic NSCLC with MET Exon 14 skipping mutation and brain metastases (BM) who received treatment with capmatinib in real-world practice settings.

The study population consisted of patients with histologically confirmed stage IIIB, IIIC, or IV MET Exon 14 skipping mutated NSCLC with BM. The date of the initiation of therapy with capmatinib after the date of initial BM diagnosis at or after the initial advanced or metastatic NSCLC diagnosis defined the study index date. The 12-month period before the study index date defined the baseline period to assess baseline demographic and clinical characteristics. Study measures were assessed at the index and during the baseline and postindex date periods. The index date needed to occur between 1 May 2020 and the date of data abstraction, provided the selected patients meet the requirement of a minimum of 6 months follow-up time available after capmatinib initiation; the exceptions to this are those patients who died during this period.

ELIGIBILITY:
Inclusion Criteria

* Patient was aged ≥ 18 years at the time of NSCLC diagnosis
* Patient had histologically confirmed stage IIIB, IIIC, or IV NSCLC with MET Exon 14 skipping mutation at the time of initial NSCLC diagnosis
* Patient had ≥ 1 measurable intracranial lesion after initial diagnosis of BM
* Patient was treated with capmatinib after diagnosis of BM (any line)

Exclusion Criteria

* Patients with characterized Epidermal Growth Factor Receptor (EGFR) and Anaplastic Lymphoma Kinase (ALK) mutations that predict sensitivity to epidermal growth factor receptor therapy, including but not limited to exon 19 deletions and exon 21 mutations
* Patients with other known actionable molecular alterations (such as ROS1 translocation or BRAF mutation) who might be candidates to receive alternative targeted therapies
* Patients who had been treated with METis in any therapy line before or after the study index date
* Patients who had participated in a clinical trial related to treatment for NSCLC at any time before or after the study index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time-to-treatment discontinuation (TTD) from treatment initiation until discontinuation of capmatinib line of therapy or death, whichever was earlier | Up to 12 months

SECONDARY OUTCOMES:
Real-world overall response rate (rwORR): Percentage of participants with best overall response of either a complete response (CR) or a partial response (PR) to the capmatinib line of therapy | Up to approximately 23 months
  rwORR was assessed per the pseudo-Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or as assessed by a healthcare professional (HCP), as available. CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions. Best overall response consisted of CR+PR.
Real-world disease control rate (rwDCR): Percentage of participants with best overall response to the capmatinib line of therapy of either CR+PR or stable disease (SD) | Up to approximately 23 months
  rwDCR was assessed per the pseudo-RECIST version 1.1 or as assessed by an HCP, as available.
Real-world duration of response (rwDOR): Time from the date of first documented CR or PR to the first documented progression or death due to any cause | Up to approximately 33 months
  CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of diameters of target lesions.
Real-world progression-free survival (rwPFS): Time from start of capmatinib therapy until the earliest of a clinically documented systemic disease progression | Up to 12 months
Overall survival (OS): Time from start of capmatinib therapy until death | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- 18 Novartis Investigative Sites in the US, East Hanover, New Jersey, United States